CLINICAL TRIAL: NCT05276427
Title: The Impact of External Factors (Brexit and Covid 19) on Retention and Turnover Among Nurses and Consultants in NHS Grampian
Brief Title: Impact of External Factors(Brexit and Covid-19) on Retention and Turnover in the NHS
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: NHS Grampian (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2-083-21
Record Dates: First submitted 2022-02-08; First posted 2022-03-11 (Actual); Last update posted 2022-03-11 (Actual); Status verified 2022-03

CONDITIONS: Impact of BREXIT & COVID 19 on Retention and Turnover on NHS
Keywords: Impact of BREXIT & COVID 19 on Retention and Turnover on NHS

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Non clinical procedure: Completion of consent form and interview session
  Interventions: Other: Non Clinical procedure

INTERVENTIONS:
Other: Non Clinical procedure — Non clinical procedure- Informed consent completion and interview session

SUMMARY:
Problems with retention and staff turnover in the health sectors of many western countries have a long history and have thus attracted research attention over the years. The National Health Service (NHS) in the United Kingdom (UK) is not immune to this problem as it is reported that the NHS as an organisation is struggling to meet staffing demands particularly with its nursing and medical workforce. One of the ways to tackle this problem has been to recruit staffs from European union countries. With the exit of UK from the EU, there are concerns on the this departure on staffing. While the UK was still coming to terms with BREXIT and its effect on the NHS, the current COVID 19 pandemic struck and has intensified workload and demands on the health sector, particularly the NHS. As a result of this, many NHS employees believe more should be done to show they are valued and appreciated for all their hard work. Turnover is already high among clinical occupations in the NHS as people leave for various reasons. It is therefore important to study the combined effect of these external factors (BREXIT and COVID 19) on turnover and retention in the NHS Grampian. It is hoped that this study will be beneficial to NHS Grampian management and policy makers as it will aid early identification of intention to leave and possibly enhance staff retention. The study will be carried out in Scotland and will be limited to NHS Grampian. Nurses and consultants who have been in employed in NHS Grampian prior to BREXIT and COVID 19 will be invited participate. Participants will voluntarily take part in a semi structured interview which may last for about 45 to 60 minutes. The project is self-funded for the award of a PhD in management studies.

ELIGIBILITY:
Inclusion Criteria:

* Must be employed in NHS Grampian prior to January 2020.
* Must be a Nurse or Consultant

Exclusion Criteria:

* Limited to Nurses and Consultants.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Nurses who have been trained in different aspects of nursing such as paediatric, neonatal, critical care, surgical, emergency care etc and consultants who have specialist training in specific aspect of medicine who have had to deal with the impact and pressures of COVID 19 and BREXIT will be invited to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2022-03 (Estimated); Primary Completion 2023-08-31 (Estimated); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
Participants will be interviewed to assess the impact of external factors on retention and turnover. | 45- 60 minutes

SECONDARY OUTCOMES:
Interviews with 40 participants will be analysed using NVivo qualitative software. | 45-60minutes

CONTACTS AND LOCATIONS:
Overall Officials: Donald Hislop, Principal Investigator — University of Aberdeen
Locations (1):
- Research and governance team, Aberdeen, United Kingdom

IPD SHARING:
Plan to Share IPD: No